CLINICAL TRIAL: NCT02273323
Title: Flow Mediated Dilation in Response to Consumption of Black Tea Versus Artificial Tea, in Non-tea Drinking Hypertensive Subjects.
Brief Title: Flow Mediated Dilation in Response to Black Tea
Acronym: T
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: REF-BEV-1376
Record Dates: First submitted 2014-10-21; First posted 2014-10-23 (Estimated); Results first posted 2017-02-15 (Actual); Last update posted 2017-02-15 (Actual); Status verified 2016-12

CONDITIONS: Vascular Function
Keywords: Flow mediated dilation; tea; blood pressure
MeSH Terms: interventions — Tea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tea (Experimental): Black tea
  Interventions: Other: Tea
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Tea — Single dose of black tea infusion containing approximately 400 mg flavonoids (expressed as gallic acid equivalents) with added sugar.
  Arms: Tea
Other: Placebo — Placebo: tea flavour, colouring and sugar
  Arms: Placebo

SUMMARY:
Research indicate that people who regularly drink tea have a reduced risk of stroke or heart disease. In a number of studies in which people that normally do not drink showed that their blood vessels function improved when the drunk tea. The current study tests whether a specific black tea improves vessel function in non-tea drinking hypertensive subjects.

DETAILED DESCRIPTION:
Epidemiological studies indicate that regular consumption of three cups of black tea per day reduces the risk of stroke or myocardial infarction. In a number of previous nutrition intervention studies tea has been shown to improve vascular function as assessed by Flow Mediated Dilation in various populations. The current confirmatory study tests a specific black tea against a placebo in a population of in non-tea drinking hypertensive subjects.

ELIGIBILITY:
Inclusion Criteria:

* Males and post menopausal (> 1 year) females, not on hormone replacement therapy
* Aged >18 and < 65 years
* Body mass index (BMI) of >=18.0 and =<35.0 kg/m2
* Hypertension as previously diagnosed by primary care or hospital physician.

  * If untreated, office BP between 140/90 mmHg and 160/100 mmHg on screening
  * If treated, a controlled blood pressure (<160/100) on stable medication for at least 4 weeks

Exclusion Criteria:

* Tea drinkers: having typically consumed > 1 cup of black tea per week.
* Current smoker or has stopped smoking less than 6 months before start of study
* Self reported alcohol intake of >21 units/week
* Established cardiovascular disease other than hypertension
* Clinically significant arrhythmia
* Diabetes mellitus
* Chronic Kidney Disease > stage 2
* 10-year cardiovascular risk equivalent to 20% or greater using the QRisk2 calculator
* Abnormality of laboratory blood tests considered clinically significant
* Any other significant intercurrent condition/disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Chowienczyk, Professor, Principal Investigator — Dept Clinical Pharmacology/CRF, St Thomas Hospital, London UK
Locations (1):
- Dept Clinical Pharmacology/CRF, St Thomas Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 53 subjects were screened between August 2014 and and October 2015
Pre-assignment Details: All 30 subjects meeting the inclusion criteria were randomised
Groups:
- Tea Then Placebo: Subjects first received a single acute dose of black tea infusion containing approximately 400 mg flavonoids (expressed as gallic acid equivalents) with added sugar. After a washout of at least 1 week, they received a single acute dose of placebo consisting of tea flavour, colouring and sugar.
- Placebo Then Tea: Subjects first received a single acute dose of placebo consisting of tea flavour, colouring and sugar. After a washout of at least 1 week, they received a single acute dose of black tea infusion containing approximately 400 mg flavonoids (expressed as gallic acid equivalents) with added sugar
Period: Overall Study
Arm/Group | Tea Then Placebo | Placebo Then Tea
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants who were randomised to either receive Tea first followed by Placebo or Placebo first followed by Tea
Arm/Group | All Study Participants
Number analyzed (Participants) | 30
Age, Continuous [Median (Full Range); unit: years] | 53 [23 to 65]
Gender [Count of Participants; unit: Participants]
  Female | 7
  Male | 23
Body Mass Index [Median (Full Range); unit: kg/m^2] | 26.3 [19.8 to 34.7]
Systolic blood pressure [Median (Full Range); unit: mmHg] | 145 [119 to 160]
Diastolic blood pressure [Median (Full Range); unit: mmHg] | 92 [67 to 102]

OUTCOME MEASURES:

1. Primary Outcome: Flow Mediated Dilation
Description: Flow mediated dilation (FMD) of the brachial artery was measured using vascular ultra sound and automated edge detection software:
  * 1 minute baseline scan to measure the baseline diameter of artery
  * 5 minutes of forearm occlusion at 250±30 mmHg, below the elbow (2-5 cm from antecubital crease)
  * 4 minutes FMD scan, which started immediately after release of occlusion Percentage FMD was calculated as the maximum increase in diameter after cuff release relative to the baseline diameter
Time Frame: Before and 2 hours after test product intake
Population: All participants who received at least one dose of each intervention and completed all study visits
Measure: Least Squares Mean (Standard Deviation); unit: percentage of change in diameter
Groups:
- Tea Beverage: Participants when they received a single dose of black tea infusion with added sugar
- Placebo Beverage: Participants when they received a single dose of placebo containing tea flavour, colouring and sugar
Arm/Group | Tea Beverage | Placebo Beverage
Number analyzed (Participants) | 30 | 30
percentage of change in diameter
  FMD before test product intake | 5.24 (2.42) | 5.02 (2.14)
  FMD two hours after test product intake | 6.05 (2.33) | 5.74 (2.66)
Statistical Analysis 1: Comparison: Tea Beverage vs Placebo Beverage; Estimated effect of tea vs placebo; Test type: Superiority or Other; p = 0.43, Mixed Models Analysis; Mean Difference (Final Values) = 0.23, 0.23% CI 2-sided [-0.37 to 0.83]

2. Secondary Outcome: Endothelium-independent Vasodilation
Description: Endothelium-independent dilation after glyceryl trinitrate defined as maximal percent increase in diameter
Time Frame: 2.5 hours after test product intake
Population: All participants who received at least one dose of each intervention and completed all study visits
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of change in diameter
Arm/Group | Tea Beverage | Placebo Beverage
Number analyzed (Participants) | 30 | 30
percentage of change in diameter | 12.1 [10.6 to 13.6] | 11.4 [9.9 to 12.9]
Statistical Analysis 1: Comparison: Tea Beverage vs Placebo Beverage; Estimated effect of tea vs. placebo; Test type: Superiority or Other; p = 0.20, Mixed Models Analysis; Subject=random factor; treatment, on/off medication, period = fixed effects; Mean Difference (Final Values) = 0.71, 95% CI 2-sided [-0.40 to 1.82]

3. Secondary Outcome: Systolic Blood Pressure Supine
Description: Systolic blood pressure measured while lying down
Time Frame: Before and 110 minutes after test product intake
Population: All participants who received at least one dose of each intervention and completed all study visits
Measure: Least Squares Mean (Standard Deviation); unit: mmHg
Arm/Group | Tea Beverage | Placebo Beverage
Number analyzed (Participants) | 30 | 30
mmHg
  Before test product intake | 135.5 (14.2) | 138.1 (14.0)
  After test product intake | 145.0 (16.2) | 147.2 (15.7)
Statistical Analysis 1: Comparison: Tea Beverage vs Placebo Beverage; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -1.35, 95% CI 2-sided [-5.26 to 2.55]

4. Secondary Outcome: Diastolic Blood Pressure Supine
Description: Diastolic blood pressure measured while lying down
Time Frame: Before and 110 minutes after test product intake
Population: All participants who received at least one dose of each intervention and completed all study visits
Measure: Least Squares Mean (Standard Deviation); unit: mmHg
Arm/Group | Tea Beverage | Placebo Beverage
Number analyzed (Participants) | 30 | 30
mmHg
  Before test product intake | 85.1 (10.2) | 85.7 (10.2)
  After test product intake | 88.9 (10.9) | 89.5 (10.5)
Statistical Analysis 1: Comparison: Tea Beverage vs Placebo Beverage; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.40, 95% CI 2-sided [-2.16 to 1.37]

5. Secondary Outcome: Systolic Blood Pressure Sitting
Description: Systolic blood pressure measured while sitting
Time Frame: Before and 90 minutes after test product intake
Population: All participants who received at least one dose of each intervention and completed all study visits
Measure: Least Squares Mean (Standard Deviation); unit: mmHg
Arm/Group | Tea Beverage | Placebo Beverage
Number analyzed (Participants) | 30 | 30
mmHg
  Before test product intake | 134.7 (13.7) | 137.2 (13.8)
  After test product intake | 146.4 (13.1) | 148.5 (15.0)
Statistical Analysis 1: Comparison: Tea Beverage vs Placebo Beverage; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -1.89, 95% CI 2-sided [-4.65 to 0.87]

6. Secondary Outcome: Diastolic Blood Pressure Sitting
Description: Diastolic blood pressure measured while sitting
Time Frame: Before and 90 minutes after test product intake
Population: All participants who received at least one dose of each intervention and completed all study visits
Measure: Least Squares Mean (Standard Deviation); unit: mmHg
Arm/Group | Tea Beverage | Placebo Beverage
Number analyzed (Participants) | 30 | 30
mmHg
  Before test product intake | 86.1 (10.3) | 87.7 (10.5)
  After test product intake | 90.7 (10.5) | 89.4 (10.0)
Statistical Analysis 1: Comparison: Tea Beverage vs Placebo Beverage; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 1.68, 95% CI 2-sided [-0.73 to 4.09]

ADVERSE EVENTS:
Arm/Group | Tea Beverage | Placebo Beverage
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 1/30 | 1/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tea Beverage (N=30) | Placebo Beverage (N=30)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days